CLINICAL TRIAL: NCT03066570
Title: Graded Exposure in Patients With Painful Diabetic Neuropathy
Acronym: PDN&GEXP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NL 57919.068.16
Record Dates: First submitted 2017-02-06; First posted 2017-02-28 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-11

CONDITIONS: Painful Diabetic Neuropathy; Diabetic Neuropathies, Painful; Neuralgia, Diabetic
Keywords: Graded Exposure; Quality of Life; Physical Activity; Anxiety
MeSH Terms: conditions — Diabetic Neuropathies; Motor Activity; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Randomized replicated sequential single-case design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single case study (Experimental): Single case study using Graded exposure.
  Interventions: Behavioral: Graded Exposure

INTERVENTIONS:
Behavioral: Graded Exposure — Graded Exposure in vivo (GEXP) is a second-generation cognitive-behavioural intervention, and is characterized by systematic and repeated exposure to feared movements, activities and/or sensations in order to decrease fear and subsequently increase physical activity.

SUMMARY:
Objective: To investigate the effects of a cognitive behavioural intervention targeting specific fears in patients with painful diabetic neuropathy, on physical activity and quality of life.

DETAILED DESCRIPTION:
Intervention: Graded Exposure in vivo (GEXP) is a second-generation cognitive-behavioural intervention, and is characterized by systematic and repeated exposure to feared movements, activities and/or sensations in order to decrease fear and subsequently increase physical activity.

Main study parameters/endpoints: The purpose of this project is to develop and test a cognitive behavioural intervention targeting specific fears in patients with PDN, in order to increase physical activity and improve QOL.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type II diabetes mellitus,
* aged > 18 years who suffer from peripheral polyneuropathy.

Exclusion Criteria:

* Patients with lower limb morbidities other than PDN such as peripheral arterial disease
* severe osteoarthritis, any other neurological disease than PDN or any other disease that may cause pain in the feet and/or damage to the peripheral nervous system (e.g. ulcers).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-03-18 (Actual); Study Completion 2019-03-18 (Actual)

PRIMARY OUTCOMES:
Quality of Life as measured with Norfolk Quality of Life Questionnaire, Diabetic Neuropathy Version (Norfolk-QOL-DN) | The primary outcome measure will be measured after 8 weeks of treatment with GEXP.
  Quality of life (QOL) will be measured using the 33-item Norfolk Quality of Life Questionnaire, Diabetic Neuropathy Version (Norfolk-QOL-DN), a self-administered questionnaire designed to capture and quantify the perceived impact of diabetic neuropathy on the QOL, physical and psychosocial functioning of patients with diabetic neuropathy.

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Geelen, MD, Study Director — charlotte.geelen@mumc.nl
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No